CLINICAL TRIAL: NCT00903695
Title: Nutriceutical Effects on Cognitive Status in Mild Cognitive Impairment Patients
Brief Title: MemoryXL Effects on Mild Cognitive Impairment Patients
Acronym: MemoryXL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Risk/benefit ratio did not indicate further study would be useful, or fair to future subjects.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14594
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Mild Cognitive Impairment
Keywords: Memory XL; Mild Cognitive Impairment; cognitive status
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memory XL (Experimental): Subjects will take 2 Memory XL pills daily for 12 months (a vitamin nutriceutical developed by Thomas Shea, Ph.D.).
  Mild Cognitive Impairment (MCI) patients, who met inclusion/exclusion criteria, were assessed initially using 3 cognitive tests and 4 behavioral questionnaires, before they began ingesting pills assigned to them by VAMC Research Pharmacist. Each 3 months thereafter, they returned to lab to be reassessed using same instruments, and to receive the next batch of study pills from the Pharmacist. The last assessment was when the patient had just finished 12 months of pill ingestion.
  Interventions: Drug: Memory XL
- placebo (Placebo Comparator): Subjects diagnosed with MCI took two placebo pills daily for 12 months; these pills are formulated to look and taste the same as the nutriceutical being studied, Memory XL, so study was double-blind. Procedures for this arm are exactly the same as the MEMORY XL arm.
  MCI subjects were assessed using 3 cognitive tests and 4 behavioral questionnaires, before they began ingesting the pills assigned to them by the Research Pharmacist at VAMC. Each 3 months thereafter, they returned to lab to be reassessed using the same instruments, and to receive next batch of study pills. Last assessment was when patient had completed 12 months of pill ingestion.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Memory XL — An over-the-counter vitamin nutriceutical patented by Univ. of Mass. that contains folic acid 400 mg, Vit. B12 6 ug, alpha-tocopherol 30 IU, S-adenosyl methionine (SAM) 400 mg, N-acetyl cysteine (NAC) 600 mg, & acetyl-L-carnitine (ALCAR) 500 mg; 2 pills per day for 12 months
  Other Names: nutriceutical
  Arms: Memory XL
Drug: placebo — placebo comparator
  Arms: placebo

SUMMARY:
A vitamin nutriceutical, Memory XL, has been shown to provide maintenance of cognitive status in mild, moderate, and severe Alzheimer's disease patients (2 publications by T. Shea). Because this nutriceutical is now patented by the Univ. of Mass., other trials at that institution may be considered a conflict of interest. Therefore, a study of its effects on Mild Cognitive Impairment (MCI) patients will be conducted by PI who is not affiliated with Univ. of Mass. or with Dr. Shea. The study hypothesis is: Memory XL will maintain or improve the cognitive and behavioral status of patients diagnosed with MCI during the year of participation in the study; normally, 10-25% of MCI patients convert to mild Alzheimer's dementia each year.

DETAILED DESCRIPTION:
This IRB-approved study is a randomized double blind study of patients diagnosed with Mild Cognitive Impairment (MCI) in the Center for Alzheimer's and Neurodegenerative Disorders (CANDO) at VAMC in Oklahoma City. Dr. Shea provided the pills (nutriceutical and placebos) from the same batches he used in former studies of Alzheimer's disease patients (produced by Nutricap Labs, Farmingdale, NY). Pills were dispensed by the OKC VAMC research pharmacist, using a random numbering system. The PI completed five cognitive testing sessions, lasting 1 to 1.5 hours, for each subject during the 12 months of participation in the study. Subject's spouse or family member completed 4 questionnaires about the subject's behavioral changes, and kept daily records of the times each day when the subject ingested the study pill assigned by the pharmacist. All subjects are patients in the VAMC memory loss clinic (CANDO) who are monitored by their neurologists (2 co-investigators in this study).

ELIGIBILITY:
Inclusion Criteria:

* MCI patients diagnosed at the VAMC Center for Alzheimers and Neurodegenerative Disorder (CANDO).
* Clinical Dementia Rating (CDR) score of 0.5.
* fluent in English.
* able to ambulate to the outpatient clinic and research laboratory
* have sight and hearing levels sufficient to complete neuropsychological testing.
* free from bipolar disorder and terminal illnesses such as cancer.
* must live with a spouse or adult relative who will record nutriceutical ingestion daily.
* subjects will be consecutively diagnosed patients from all ethnic groups.

Exclusion Criteria:

* patients from protected categories such as prisoners and pregnant women.
* any MCI subject who develops a life-threatening disease such as terminal cancer, stroke, brain trauma, debilitating heart attack, etc.
* indication of inability to make decisions regarding study participation.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilee Monnot, Ph.D., Principal Investigator — University of Oklahoma HSC
Locations (2):
- United States (2):
  - Univ. of Okla. Health Sciences Center & VAMC OKC, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center, Oklahoma City, Oklahoma

REFERENCES:
- [Background] Chan, A., Paskavitz, J., Remington, J.R., Rasmussen, S., Shea, T.B. (2009).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with Mild Cognitive Impairment (MCI) in VA and OU campus clinics were given opportunity to participate in the trial, if they met inclusion/exclusion criteria.
Pre-assignment Details: Over 1.5 yrs, only 19 of 533 memory clinic patients were diagnosed with Mild Cognitive Impairment and who met inclusion/exclusion criteria. Most of the MCI patients had serious medical problems that affected cognition. Ten subjects agreed to be in this study.
Groups:
- Nutriceutical (MemoryXL) Effects on Cognition & Behavior: Subjects diagnosed with Mild Cognitive Impairment (MCI) will take 2 Memory XL pills daily for 12 months (a vitamin nutriceutical developed by Thomas Shea, Ph.D., and patented by the Univ. of Mass.). They will be assessed cognitively each 3 months to determine if Memory XL prevents them from progressing to early dementia; 10-25% of MCI patients have been shown to convert to dementia each year. Therefore, at least 10% of patients in study would be expected to progress from MCI to early Alzheimer's dementia during the year of the study.
- Placebo Effects on Cognition/Behavior: Mild Cognitive Impairment subjects will take the placebo that has been formulated to look and taste the same as the nutriceutical being studied (Memory XL). Subjects will be cognitively & behaviorally assessed each 3 months of the study, with last testing done at the end of their 12 months of pill ingestion. Tests used in each arm of study are the same ones used in prior publications by the nutriceutical inventor, Dr. Shea, when he assessed mild, moderate, and severely demented Alzheimer's patients. The current study is double blind, whereas Dr. Shea's studies were open label.
Period: Overall Study
Arm/Group | Nutriceutical (MemoryXL) Effects on Cognition & Behavior | Placebo Effects on Cognition/Behavior
Started | 8 | 2
Completed | 6 | 2
Not Completed | 2 | 0
Not completed — medical exclusion after 1st testing | 1 | 0
Not completed — lung cancer | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nutriceutical (MemoryXL) Effects on Cognition & Behavior | Placebo Effects on Cognition/Behavior | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 2 | 10
Dementia Rating Scale [Mean (Standard Deviation); unit: total raw score points for 5 domains] — Dementia Rating Scale (DRS) = cognitive test with 5 domains; raw scores can be converted to percentiles for age/education levels. Higher scores mean more competence (range = 0 to 180 points).
  total raw score points for 5 domains | 130 (2.3) | 140 (4.7) | 132 (7.5)
MiniMental State Exam (MMSE) [Mean (Standard Deviation); unit: total 1st MMSE score parameters] — MiniMental State Exam (MMSE) is a cognitive screening device with possible 30 points; higher scores mean more competence, and scores can range from 0-30 points.
  total 1st MMSE score parameters | 27.5 (0.8) | 28.5 (1.5) | 27.7 (2.1)
Neuropsychiatric Inventory NPI) [Mean (Standard Deviation); unit: total raw scores by group] — Neuropsychiatric Inventory (NPI) behavior rating scale includes 12 domains; higher numbers mean more psychiatric pathology (0 to 36 points).
  total raw scores by group | 3.6 (1.3) | 3.0 (2.6) | 3.5 (3.4)
Modified Clinical Dementia Rating scale (CDR) [Mean (Standard Deviation); unit: total raw scores by study group] — Modified CDR is a behavior rating scale of 8 domains, with 5 incremental scores for each domain (0, 0.5, 1, 2, 3). Total raw score of 0 means patient is healthy; raw score of 1 to <8 points from the 8 domains earns subject a CDR scale score of 0.5 (Mild Cognitive Impairment, no dementia). Total scaled score of 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia.
  total raw scores by study group | 5.6 (1.4) | 6.5 (2.8) | 5.8 (3.8)
Activities of Daily Living (ADL) [Mean (Standard Deviation); unit: total initial raw scores by group] — ADL is a behavior rating scale with 6 domains of self-care (feeding, toileting, etc.), with 3 incremental scores (1, 2, 3) in which higher scores mean more pathology (total scores of 6 to 18 points).
  total initial raw scores by group | 6.3 (0.4) | 8.0 (0.7) | 6.6 (1.2)
Instrumental Activities of Daily Living (IADL) [Mean (Standard Deviation); unit: total initial scores by study group] — IADL is a behavior rating scale with 9 domains, and 3 incremental scores ( 1, 2, 3). Total scores can range from 9 to 27, with higher scores indicating more pathology.
  total initial scores by study group | 14.2 (1.8) | 13.0 (3.7) | 14.0 (4.9)
Clock Drawing Test [Mean (Standard Deviation); unit: initial total raw score by group] — Clock Drawing Test is a cognitive screening instrument in which subjects are asked to draw a traditional clock and place the hands at a specified time. Scoring in this version used 8 indicators of accuracy and skill, with higher scores showing more competence (0-8 pts possible).
  initial total raw score by group | 6.7 (0.3) | 7.0 (0.7) | 6.8 (0.9)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Subjects Who Converted to Early Alzheimer's (Dementia).
Description: Neurological diagnosis is based on test scores that reach -1.6 SD of mean for age/education, and on radiological tests of brain structure (CT, MRI, PET). Usual cutoff for test score percentile is <0.05 to diagnose dementia.
Time Frame: 12 months
Population: Subjects diagnosed as Mild Cognitive Impairment (MCI) in VA clinic were given opportunity to participate in the study if they met inclusion/exclusion criteria (no illnesses that cause brain damage or are uncontrolled such as brittle diabetes).
Measure: Number; unit: participants
Groups:
- Nutriceutical Arm: Subjects who were assigned by VA research pharmacist to receive nutriceutical pills for full 12 months of study. They were told to take one pill each in AM and PM, and spouse kept a log of the time of day when subject injected the pill. Logs were brought to PI each three months when patient returned to lab for re-testing and to receive next batch of study pills.
- Placebo Arm: Subjects who were assigned by VA research pharmacist to receive placebo pills for full 12 months of study. They were told to take one pill each in AM and PM, and spouse kept a log of the time of day when subject injected the pill. Logs were brought to PI each three months when patient returned to lab for re-testing and to receive next batch of study pills.
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
participants | 0 | 1

2. Primary Outcome: Differences in Dementia Rating Scale (DRS) at 12 Months From Baseline, by Study Group
Description: Dementia Rating Scale (DRS) is a cognitive test with 5 domains; raw scores can be converted to percentiles for age/education levels, so individuals can be compared. Higher scores mean more competence (0-36 points converted to percentiles so different ages can be compared). Total raw scores for the 5 domains were computed so that Mean and SD of differences between first and last assessments for all subjects, by study arms (nutriceutical = XL and placebo = PL) are reported here.
Time Frame: Baseline and 12 months
Population: All participants who completed 12-month study were included in the ANOVA analysis of the differences in scores of tests between baseline and end assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nutriceutical (MemoryXL) Effects on Cognition & Behavior | Placebo Effects on Cognition/Behavior
Number analyzed (Participants) | 6 | 2
units on a scale | -1.0 (3.0) | -2.5 (5.3)
Statistical Analysis 1: Comparison: Nutriceutical (MemoryXL) Effects on Cognition & Behavior vs Placebo Effects on Cognition/Behavior; ANOVA used to detect significant difference in test scores between baseline and end assessments, by study arm (nutriceutical vs placebo); Test type: Superiority or Other; p = 0.8133, ANOVA — a priori threshold for statistical significance = 0.01 (multiple comparisons); DF = 6 ANOVA calculation: F-ratio = 0.06, t-test = -0.25

3. Primary Outcome: Differences in Clinical Dementia Rating Scale (CDR) Over 12 Months, by Study Group
Description: CDR is a rating scale for 8 aspects of behavior with 0-3 points allowed; higher scores indicate more pathology. Total minimum and maximum scores are 0 and 36 respectively.Clinician rates the patient's behavior and competence with input from family members who live with the patient. ANOVA of differences between baseline and end scores of the CDR scale are reported here, by the study arm/group.
Time Frame: baseline before intervention to 12 months of intervention
Population: All subjects who completed the 12-month study were included (placebo and nutriceutical arms/groups).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
units on a scale | -1.7 (1.6) | 2.0 (2.9)
Statistical Analysis 1: Comparison: Nutriceutical Arm vs Placebo Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.31, ANOVA — a priori threshold for statistical sginficance = 0.01 (multiple comparisons); DF = 6 ANOVA calculation: F-ratio=1.22, t-test=1.1

4. Primary Outcome: Differences in Clock Drawing Test (CLOX) Scores Over 12 Months, by Study Group
Description: Clock Drawing Test is a cognitive screening instrument in which subjects are to draw a clock and set a specified time. Various scoring methods can be employed using 4 to 15 points, with more points showing more competence. This study used the 8-point scoring method, so that 0-8 points could be assigned during each of the baseline and 4 assessment periods during the 12-month study. ANOVA of the differences between baseline and end scores, by study arm/group was completed.
Time Frame: baseline to 12 months
Population: All subjects who completed the 12-month study were included.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
units on a scale | 0.5 (0.6) | -1.0 (1.1)
Statistical Analysis 1: Comparison: Nutriceutical Arm vs Placebo Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.27, ANOVA — a priori threshold for statistical significance = 0.01 (multiple comparisons); DF = 6 ANOVA: F-ratio = 1.5, t-test = -1.23

5. Primary Outcome: Differences in MiniMental State Exam (MMSE) Scores Over 12 Months, by Study Group
Description: MiniMental State Exam is a cognitive screening device with possible 30 points in several categories; higher points indicate greater competence. Clinician tests orientation, attention, language, & visuo-spatial construction. Outcome measure is results of an ANOVA of differences between baseline and end/last scores, by study arm/group was completed.
Time Frame: baseline to 12 months
Population: All subjects who completed the 12-month study were included.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
units on a scale | -0.33 (0.5) | 1.0 (0.9)
Statistical Analysis 1: Comparison: Nutriceutical Arm vs Placebo Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.24, ANOVA — a priori threshold for statistical significance = 0.01 (multiple comparisons); DF = 6 ANOVA: F-ratio = 1.7, t-test = 1.3

6. Primary Outcome: Differences in Neuropsychiatric Inventory (NPI) Scores Over 12 Months, by Study Group
Description: NPI is a behavior rating scale with 12 categories in which a maximum score of 36 points indicates more pathology than a minimum score of 0. Outcome measure reported here is results of an ANOVA of the differences between baseline and end scores, by study arm/group, to detect any statistically significant difference (nutriceutical vs placebo groups) was completed.
Time Frame: baseline to 12 months
Population: All subjects who completed 12-month study were included.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
units on a scale | -4.0 (1.9) | -2.5 (3.3)
Statistical Analysis 1: Comparison: Nutriceutical Arm vs Placebo Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.71, ANOVA — a priori threshold for statistical significance = 0.01 (multiple comparisons); DF = 6 ANOVA: F-ratio = 0.15, t-test = 0.39

7. Primary Outcome: Differences in Activities of Daily Living (ADL) Scores Over 12 Months, by Study Group
Description: ADL is a behavior rating scale with 6 domains of self-care (feeding, toileting, etc.) in which a maximum score of 18 indicates less competence than a minimum score of 6 (normal skills). Outcome measure is results of ANOVA of the differences between baseline and last/end scores, by study arm/group, to detect any statistically significant differences.
Time Frame: baseline to 12 months
Population: All subjects who completed 12-month study were included.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
units on a scale | 0.0 (0.3) | -1.0 (0.6)
Statistical Analysis 1: Comparison: Nutriceutical Arm vs Placebo Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.18, ANOVA — a priori threshold for statistical significance = 0.01 (multiple comparisons); DF = 6 ANOVA: F-ratio = 2.25, ttest = -1.5

8. Primary Outcome: Differences in Instrumental Activities of Daily Living (IADL) Scores Over 12 Months, by Study Group
Description: IADL is a behavior rating scale using 9 domains of household and community activities, with a total score of 27 points indicating less competence than a normal function score of 9 points. Outcome measure is results of an ANOVA of the differences between baseline and end/last score, by study arm/group, to detect statistically significant differences (nutriceutical vs placebo).
Time Frame: baseline to 12 months
Population: All subjects who completed 12-month study were included.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nutriceutical Arm | Placebo Arm
Number analyzed (Participants) | 6 | 2
units on a scale | 0.0 (1.0) | -2.0 (1.7)
Statistical Analysis 1: Comparison: Nutriceutical Arm vs Placebo Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.34, ANOVA — a priori threshold for statistical significance = 0.01 (multiple comparisons); DF = 6 ANOVA: F-ratio = 1.06, t-test = -1.03

ADVERSE EVENTS:
Time Frame: 12-month study (double-blind) of Mild Cognitive Impairment patients recruited from VAMC Neurosciences memory loss clinic.
Arm/Group | Nutriceutical (MemoryXL) Effects on Cognition & Behavior | Placebo Effects on Cognition/Behavior
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 0/8 | 0/2

LIMITATIONS AND CAVEATS:
Benefits of study did not appear to outweigh subject inconvenience, so study was stopped prematurely. Also, very few 'healthy' MCI subjects were recruited from the clinic population; vast majority of MCI patients had exclusionary medical problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No